CLINICAL TRIAL: NCT03036657
Title: Local Effects of Acupuncture on the Median and Ulnar Nerves in Patients With Carpal Tunnel Syndrome
Brief Title: Local Effects of Acupuncture and Nerve Conduction Studies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Alexandra Dimitrova, Assistant Professor of Neurology, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRB00008949
Record Dates: First submitted 2016-08-14; First posted 2017-01-30 (Estimated); Results first posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Acupuncture; Electroacupuncture; Nerve Conduction Studies; Quantitative Sensory Testing
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Manual Acupuncture (Experimental): Device:
  Sterile single-use MAC acupuncture needles - 0.22 x 25 mm, TianJin Haing Lim Sou Won Medical Equipment Co, Ltd, South Korea
  Used for Intervention:
  Manual Acupuncture to PC3, PC5 or HT3, HT4 for 20 min
  Interventions: Device: MAC acupuncture needles
- Low-Frequency Electroacupuncture (Experimental): Device:
  Electrostimulator 6c.Pro, Pantheon Research, Venice, CA
  Used for Intervention:
  Low-frequency Continuous Electroacupuncture (2Hz) to PC3, PC5 or HT3, HT4 for 20 min
  Interventions: Device: Electrostimulator 6c.Pro, Pantheon Research, Venice, CA
- High-Frequency Electroacupuncture (Experimental): Device:
  Electrostimulator 6c.Pro, Pantheon Research, Venice, CA
  Used for Intervention:
  High-frequency Continuous Electroacupuncture (100 Hz) to PC3, PC5 or HT3, HT4 for 20 min
  Interventions: Device: Electrostimulator 6c.Pro, Pantheon Research, Venice, CA

INTERVENTIONS:
Device: MAC acupuncture needles — Sterile single-use MAC acupuncture needles (0.22 x 25 mm, TianJin Haing Lim Sou Won Medical Equipment Co, Ltd, South Korea. Used for Manual Acupuncture
  Used for: Manual Acupuncture to PC3, PC5 or HT3, HT4 for 20 min
  Arms: Manual Acupuncture
Device: Electrostimulator 6c.Pro, Pantheon Research, Venice, CA — Electrostimulator used for delivery or Low-Frequency or High-Frequency Electroacupuncture
  Used for Interventions:
  Low-frequency Continuous Electroacupuncture to PC3, PC5 or HT3, HT4 for 20 min AND High-frequency Continuous Electroacupuncture to PC3, PC5 or HT3, HT4 for 20 min
  Arms: High-Frequency Electroacupuncture; Low-Frequency Electroacupuncture

SUMMARY:
Thus study aims to characterize the local, nerve-specific effects of acupuncture on the median and ulnar nerves in the forearm, using nerve conduction studies and quantitative sensory testing. All participant will have carpal tunnel syndrome and the affected median nerve will be compared to the healthy ulnar nerve. Additionally, we aim to compare the local, nerve-specific effect of manual acupuncture to that of low-frequency electroacupuncture and of high-frequency electroacupuncture.

DETAILED DESCRIPTION:
The purpose of this study is to measure the local effects of acupuncture on the median and ulnar nerves in patients with median neuropathy at the wrist (carpal tunnel syndrome), using nerve conduction studies (NCS) and quantitative sensory testing (QST) as outcomes. Our secondary aim is to compare acupuncture's effect on the functioning of a diseased nerve (median nerve in CTS) to its effect on a healthy nerve (ulnar). Additionally, we aim to compare the local, nerve-specific effect of manual acupuncture to that of low-frequency electroacupuncture and of high-frequency electroacupuncture.

In a mechanistic study of acupuncture, 60 subjects with carpal tunnel syndrome (CTS) will be randomized to manual acupuncture (MA), low-frequency electroacupuncture (LF-EA) and high-frequency electroacupuncture (HF-EA) groups. Baseline measurements will consist of QST (vibration and cold detection thresholds), as well as NCS of both median and ulnar nerves. Then, each group will undergo acupuncture to the median nerve (Pericardium channel points) and to the ulnar nerve (Heart channel points), one week apart, order counterbalanced, followed by post-acupuncture NCS and QST measurements in both nerves' territories.

ELIGIBILITY:
Inclusion Criteria:

* Presence of mild-moderate sensorimotor or sensory median neuropathy, established by pre-existing NCS/EMG study AND
* Baseline NCS study within the past 2 years, consistent with mild-moderate median entrapment neuropathy (CTS) defined as meeting any of the 3 conditions below:

  1. Prolonged distal Median sensory AND/OR motor latency
  2. Reduced Median sensory nerve action potentials (SNAP) amplitude by no more than 50%
  3. Amplitude of the compound muscle action potential (CMAP) recorded from APB > 50% of normal
* Presence of neuropathy symptoms consistent with CTS for at least 3 months

Exclusion Criteria:

Conditions in which acupuncture/electroacupuncture may be contraindicated:

* Coagulopathy/ Current anti-coagulation treatment
* Epilepsy
* History of CAD or pacemaker insertion
* Pregnancy
* Presence of any skin condition in the arm, such as dermatitis, bruises, weeping skin, skin lesions, infected skin, or necrotic skin.

Conditions in which QST testing may be contraindicated:

* Significant cognitive impairment such as diagnosis of Alzheimer's disease or Mental Retardation or any other condition interfering with alertness, attention and ability to participate in QST
* Hospitalization for anxiety or depression in the past 3 months
* Current psychiatric diagnoses (other than anxiety or depression)
* Illicit drug use in the past month
* Current EtOH abuse (> 2 drinks/day)
* History of significant neurological disease which may affect sensation, e.g., strokes, Multiple Sclerosis, or spinal cord disorder
* Change in neuropathy medications within the past 2 months
* Change in opioid, benzodiazepines, SSRIs or other sedating medications in the past 2 months

Conditions, which predispose to generalized neuropathy

* Abnormal thyroid function tests (by history)
* Past chemotherapy treatment

Other Contraindications:

* History of wrist or elbow fracture, past arm trauma, loss of fingers, scarring
* History of carpal tunnel release surgery or any other surgery on the arm or shoulder
* History of arthritis
* Use of any investigational drugs within the previous six months

Exclusion Criteria based on NCS within the past 2 years:

* Presence of isolated motor Median neuropathy (absence of sensory neuropathy on NCS or absence of sensory symptoms)
* Severe neuropathy symptoms leading to inability to tolerate acupuncture or QST
* Presence of Severe Carpal Tunnel Syndrome, defined as:

  1. Absent sensory nerve action potential recorded from the second or fifth digit.
  2. The amplitude of the compound muscle action potential recorded from the APB or ADM is less than 50% of normal (< 2.5 mv)
* Presence of Ulnar neuropathy
* Presence of Martin-Gruber anastomosis

Secondary Exclusion Criteria after WEEK 1 Baseline QST and NCS measurements:

* Failure to comply with QST due to inattentiveness, etc
* Hyperalgesia on QST
* Hypoalgesia on QST
* Inability to confirm diagnosis of mild-moderate CTS (normal NCS)
* Inability to tolerate NCS/QST
* Presence Severe CTS
* Pure Motor Median Neuropathy
* Ulnar Neuropathy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-10; Primary Completion 2021-05 (Actual); Study Completion 2021-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Derived] Dimitrova A, Murchison C, Oken B. Local effects of acupuncture on the median and ulnar nerves in patients with carpal tunnel syndrome: a pilot mechanistic study protocol. Trials. 2019 Jan 5;20(1):8. doi: 10.1186/s13063-018-3094-5. PMID 30611294

RESULTS

PARTICIPANT FLOW:
Groups:
- Manual Acupuncture: Device:
  Sterile single-use MAC acupuncture needles - 0.22 x 25 mm, TianJin Haing Lim Sou Won Medical Equipment Co, Ltd, South Korea
  Used for Intervention:
  Manual Acupuncture to PC3, PC5 or HT3, HT4 for 20 min
  MAC acupuncture needles: Sterile single-use MAC acupuncture needles (0.22 x 25 mm, TianJin Haing Lim Sou Won Medical Equipment Co, Ltd, South Korea. Used for Manual Acupuncture
  Used for: Manual Acupuncture to PC3, PC5 or HT3, HT4 for 20 min
- Low-Frequency Electroacupuncture: Device:
  Electrostimulator 6c.Pro, Pantheon Research, Venice, CA
  Used for Intervention:
  Low-frequency Continuous Electroacupuncture (2Hz) to PC3, PC5 or HT3, HT4 for 20 min
  Electrostimulator 6c.Pro, Pantheon Research, Venice, CA: Electrostimulator used for delivery or Low-Frequency or High-Frequency Electroacupuncture
  Used for Interventions:
  Low-frequency Continuous Electroacupuncture - 4 Hz to PC3, PC5 or HT3, HT4 for 20 min AND
- High-Frequency Electroacupuncture: Device:
  Electrostimulator 6c.Pro, Pantheon Research, Venice, CA
  Used for Intervention:
  High-frequency Continuous Electroacupuncture (100 Hz) to PC3, PC5 or HT3, HT4 for 20 min
  Electrostimulator 6c.Pro, Pantheon Research, Venice, CA: Electrostimulator used for delivery or Low-Frequency or High-Frequency Electroacupuncture
  Used for Interventions:
  High-frequency Continuous Electroacupuncture - 100 Hz to PC3, PC5 or HT3, HT4 for 20 min
Period: Overall Study
Arm/Group | Manual Acupuncture | Low-Frequency Electroacupuncture | High-Frequency Electroacupuncture
Started | 20 | 20 | 20
Completed | 20 | 20 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Low-Frequency Electroacupuncture: Device:
  Electrostimulator 6c.Pro, Pantheon Research, Venice, CA
  Used for Intervention:
  Low-frequency Continuous Electroacupuncture (2Hz) to PC3, PC5 or HT3, HT4 for 20 min
  Electrostimulator 6c.Pro, Pantheon Research, Venice, CA: Electrostimulator used for delivery or Low-Frequency or High-Frequency Electroacupuncture
  Used for Interventions:
  Low-frequency Continuous Electroacupuncture to PC3, PC5 or HT3, HT4 for 20 min AND High-frequency Continuous Electroacupuncture to PC3, PC5 or HT3, HT4 for 20 min
- High-Frequency Electroacupuncture: Device:
  Electrostimulator 6c.Pro, Pantheon Research, Venice, CA
  Used for Intervention:
  High-frequency Continuous Electroacupuncture (100 Hz) to PC3, PC5 or HT3, HT4 for 20 min
  Electrostimulator 6c.Pro, Pantheon Research, Venice, CA: Electrostimulator used for delivery or Low-Frequency or High-Frequency Electroacupuncture
  Used for Interventions:
  Low-frequency Continuous Electroacupuncture to PC3, PC5 or HT3, HT4 for 20 min AND High-frequency Continuous Electroacupuncture to PC3, PC5 or HT3, HT4 for 20 min
- Total: Total of all reporting groups
Arm/Group | Manual Acupuncture | Low-Frequency Electroacupuncture | High-Frequency Electroacupuncture | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 17 | 16 | 15 | 48
  >=65 years | 3 | 4 | 5 | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.05 (13.33) | 48.90 (17.22) | 55.50 (13.92) | 52.15 (14.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 16 | 48
  Male | 4 | 4 | 4 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 19 | 19 | 20 | 58
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 19 | 19 | 18 | 56
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 20 | 60
Median Cold Detection Threshold [Mean (Standard Deviation); unit: JND (just noticeable difference)] | 8.0 (2.3) | 8.6 (1.9) | 7.8 (1.6) | 8.2 (1.9)
Ulnar Cold Detection Threshold [Mean (Standard Deviation); unit: JND (Just Noticeable Difference)] | 10.1 (2.2) | 10.8 (2.3) | 10.2 (2.0) | 10.4 (2.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Median Cold Detection Threshold (CDT) Post-acupuncture Compared to Pre-acupuncture When the Median Nerve is Treated
Description: The median change plus standard deviation when the median nerve was treated and CDT was measured in the sensory distribution of the median nerve.
  The CDT is measured in CASE IV - specific units named Just Noticeable Difference (JND). The CASE IV System uses a set of 25 standardized vibratory and thermal stimulation levels for patient testing and analysis. These 25 levels are termed "Just Noticeable Differences" or "JNDs," and are similar to decibels. The concept of a JND is based on the fact that a sensitive person can detect fine differences between two levels of stimulation, whereas an insensitive person cannot. Because differences of less than one JND are difficult to distinguish, one JND is the smallest difference presented to patients. Stimuli based on the JND scale can be used to test patients very efficiently and quickly, without compromising the significance of the clinical result.
Time Frame: Week 1, Week 2
Measure: Median (Standard Deviation); unit: JND (just noticeable difference)
Arm/Group | Manual Acupuncture | Low-Frequency Electroacupuncture | High-Frequency Electroacupuncture
Number analyzed (Participants) | 20 | 20 | 20
JND (just noticeable difference) | 0.73 (1.527) | -0.195 (1.698) | 0.865 (2.021)

2. Primary Outcome: Change in Ulnar Cold Detection Threshold (CDT) Post-acupuncture Compared to Pre-acupuncture When the Median Nerve is Treated
Description: This is the mean change plus standard deviation in CDT in the sensory distribution of the ulnar never when the median nerve is treated.
  The CDT is measured in CASE IV - specific units named Just Noticeable Difference (JND). The CASE IV System uses a set of 25 standardized vibratory and thermal stimulation levels for patient testing and analysis. These 25 levels are termed "Just Noticeable Differences" or "JNDs," and are similar to decibels. The concept of a JND is based on the fact that a sensitive person can detect fine differences between two levels of stimulation, whereas an insensitive person cannot. Because differences of less than one JND are difficult to distinguish, one JND is the smallest difference presented to patients. Stimuli based on the JND scale can be used to test patients very efficiently and quickly, without compromising the significance of the clinical result.
Time Frame: Week 1, Week 2
Measure: Mean (Standard Deviation); unit: JND
Arm/Group | Manual Acupuncture | Low-Frequency Electroacupuncture | High-Frequency Electroacupuncture
Number analyzed (Participants) | 20 | 20 | 20
JND | 0.215 (1.732) | 0.07 (1.264) | 0.375 (1.064)

3. Primary Outcome: Change in Median Cold Detection Threshold (CDT) Post-acupuncture Compared to Pre-acupuncture When the Ulnar Nerve is Treated
Description: This is the mean change plus standard deviation in the sensory territory of the Median nerve when the Ulnar nerve was treated.
Time Frame: Week 1, Week 2
Measure: Mean (Standard Deviation); unit: JND
Arm/Group | Manual Acupuncture | Low-Frequency Electroacupuncture | High-Frequency Electroacupuncture
Number analyzed (Participants) | 20 | 20 | 20
JND | -0.37 (1.309) | 0.23 (1.358) | 0.23 (1.627)

4. Primary Outcome: Change in Ulnar Cold Detection Threshold (CDT) Post-acupuncture Compared to Pre-acupuncture When the Ulnar Nerve is Treated
Description: This is the mean plus standard deviation change in CDT in the sensory territory of the ulnar nerve when the ulnar nerve is treated.
Time Frame: Week 1, Week 2
Measure: Mean (Standard Deviation); unit: JND
Arm/Group | Manual Acupuncture | Low-Frequency Electroacupuncture | High-Frequency Electroacupuncture
Number analyzed (Participants) | 20 | 20 | 20
JND | -0.68 (1.626) | 0.30 (1.182) | 0.405 (0.990)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the period of study enrollment, which ended after completion of visit #2 at week #2. In addition, participants were encouraged to contact the PI and the IRB with any issues of concerns after exiting the study.
Description: Risk for SAEx was minimal. The study was minimally invasive, consisted placement of 2 acupuncture needles in the forearm per visit.
  The risk for all-cause Mortality was negligible due to the exclusion criteria eliminating multiple serious pre-existing conditions.
  The number of participants at risk of unanticipated adverse events was negligible as the study was considered minimally invasive.
Arm/Group | Manual Acupuncture | Low-Frequency Electroacupuncture | High-Frequency Electroacupuncture
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2015-07-27): https://cdn.clinicaltrials.gov/large-docs/57/NCT03036657/Prot_SAP_ICF_000.pdf